CLINICAL TRIAL: NCT01058811
Title: Established Lung Cancer Cell Line and Stroma Cell From Surgical Tissue: Find Lung Cancer Stem Cells and Test Its Chemotherapy Drug Resistance; Compare Stroma Cell Between Tumor Part and Surrounding Part
Brief Title: Established Lung Cancer Cell Line and Stroma Cell From Surgical Tissue
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Department of Health, Executive Yuan, R.O.C. (Taiwan) (Other Government); National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Chao-Chi Ho, National Taiwan University Hospital
Other Study IDs: 200912012R
Record Dates: First submitted 2010-01-27; First posted 2010-01-29 (Estimated); Last update posted 2010-01-29 (Estimated); Status verified 2010-01

CONDITIONS: Lung Cancer
Keywords: lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Routine Surgical resection of lung tumor
Oversight: Data Monitoring Committee: No

SUMMARY:
Try to find lung cancer stem cells from primary culture of routine surgical resection of lung cancer tissue including cancer cells and stroma cells, then characterization the established cell lines, and compare the difference of stroma cells between tumor part and surrounding part.

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patient with surgical resection of lung tumor

Exclusion Criteria:

* lung cancer patient without surgical resection of lung tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: lung cancer patient
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2009-12; Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chi Ho, MD PhD, Study Chair — National Taiwan University Hospital, Taipei, Taiwan
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan